CLINICAL TRIAL: NCT05970016
Title: A Phase I/II Clinical Study to Evaluate the Tolerability, Safety, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of TCC1727 Tablets in Patients with Advanced Solid Tumor.
Brief Title: A Phase I/II Clinical Study in Patients with Advanced Solid Tumor.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Tide Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCC1727-101
Record Dates: First submitted 2023-07-14; First posted 2023-08-01 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Patients with Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (11):
- 5mg treatment group (Experimental): Administered orally once a day (QD)
  Interventions: Drug: TCC1727 tablet（1）
- 10mg treatment group (Experimental): Administered orally once a day (QD)
  Interventions: Drug: TCC1727 tablet（1）
- 20mg treatment group (Experimental): Administered orally once a day (QD)
  Interventions: Drug: TCC1727 tablet（1）
- 40mg treatment group (Experimental): Administered orally once a day (QD)
  Interventions: Drug: TCC1727 tablet（1）
- 60mg treatment group (Experimental): Administered orally once a day (QD)
  Interventions: Drug: TCC1727 tablet（1）
- 80mg treatment group (Experimental): Administered orally once a day (QD)
  Interventions: Drug: TCC1727 tablet（1）
- 100mg treatment group (Experimental): Administered orally once a day (QD)
  Interventions: Drug: TCC1727 tablet（1）
- 60mg BID treatment group (Experimental): Drug: TCC1727 tablet TCC1727 tablet will be administered orally twice a day (BID) every morning , and 21 days/cycle on an empty stomach.
  Interventions: Drug: TCC1727 tablet（2）
- 90mg BID treatment group (Experimental): Drug: TCC1727 tablet TCC1727 tablet will be administered orally twice a day (BID) every morning, and 21 days/cycle on an empty stomach.
  Interventions: Drug: TCC1727 tablet（2）
- 120mg BID treatment group (Experimental): Drug: TCC1727 tablet TCC1727 tablet will be administered orally twice a day (BID) every morning, and 21 days/cycle on an empty stomach.
  Interventions: Drug: TCC1727 tablet（2）
- 160mg BID treatment group (Experimental): Drug: TCC1727 tablet TCC1727 tablet will be administered orally twice a day (BID) every morning, and 21 days/cycle on an empty stomach.
  Interventions: Drug: TCC1727 tablet（2）

INTERVENTIONS:
Drug: TCC1727 tablet（1） — TCC1727 tablet will be administered orally once a day (QD) every morning for 3 days followed by discontinuation for 4 days, and 21 days/cycle on an empty stomach.
  Arms: 100mg treatment group; 10mg treatment group; 20mg treatment group; 40mg treatment group; 5mg treatment group; 60mg treatment group; 80mg treatment group
Drug: TCC1727 tablet（2） — Drug: TCC1727 tablet TCC1727 tablet will be administered orally twice a day (BID) every morning , and 21 days/cycle on an empty stomach.
  Arms: 120mg BID treatment group; 160mg BID treatment group; 60mg BID treatment group; 90mg BID treatment group

SUMMARY:
This is a 2-part, phase I/II, open-label, multicenter study designed to evaluate the safety, PK, PD and preliminary efficacy of TCC1727 tablets administered orally QD.

DETAILED DESCRIPTION:
The study will be divided into two stages: the first stage is a phase I dose finding study in patients with advanced solid tumors; the second stage is a phase II cohort expansion study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects who have provided voluntary informed consent for participation in the study and to follow the protocol requirements
2. Male or female subjects 18-70 years of age
3. Subjects with histologically or cytologically confirmed malignant advanced solid tumors who have progressed on (or have not been able to tolerate) standard therapy or for whom no suitable effective standard therapy exists

   1. For Phase I, all tumor types will be enrolled
   2. For Phase II, Patients with DDR defects detection at central laboratory will be enrolled
4. Subject with at least one measurable lesion according to RECIST criteria (version 1.1) for solid tumors will be allowed to include in phase II (if there is no measurable lesion but there are assessable lesions then the subject will be allowed to be included after the judgment of the investigator in phase I only)
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Subjects with life expectancy of ≥12 weeks
7. Subjects 12-lead ECG evaluation of QT level using Fridericia formula (QTcF) < 450 mse
8. Subjects must have the following laboratory values:

   1. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L;
   2. Platelet count (PLT) ≥ 100 × 109/L;
   3. Hemoglobin (HB) ≥ 9.0 g/L;
   4. No blood transfusion or hematopoietic stimulating factor treatment within 14 days;
   5. Bilirubin total ≤ 1.5 times the upper limit of normal (ULN);
   6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN (In case of liver metastasis, ALT and AST ≤ 5 × ULN);
   7. 24-hour or calculated creatinine clearance (CrCl) ≥ 60 mL/min (according to Cockcroft-Gault formula)*, or the 24-hour creatinine clearance measured in urine is ≥ 50 mL/min, the patient will still be selected. *For CrCl value, the eligibility should be determined using the Cockcroft-Gault formula:

      * Male CrCl (mL/min) = body weight (kg) × (140 - age)/[72 × serum creatinine (mg/dL)]
      * Female CrCl (mL/min) = male CrCl × 0.85
   8. International normalized ratio (INR) ≤ 1.5 × ULN, Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN;
9. Women of childbearing potential agreed to use effective contraceptives during the study treatment period and within 3 months after the end of the study treatment period.

Exclusion Criteria:

Subjects will be excluded from the study based on the following criteria:

1. Imaging examination suggests intracranial metastasis, which requires local treatment (in case of asymptomatic or symptomatic brain metastasis requiring no local treatment based on the investigator's judgement, the subject can still be included), or currently taking steroid hormone prior to inclusion, such as >10 mg prednisone (or equivalent) for intracerebral edema from brain metastases; subjects with meningeal carcinomatosis will be excluded regardless of their clinical stability
2. History of previously received major surgery or surgical therapy for any cause within 4 weeks of the first dose; radiotherapy, chemotherapy, other clinical trial drugs or other anti-tumor treatment, within 5 half-lives or 3 weeks (whichever is shorter), prior administering the first dose of study drug on Day 1
3. History of previous treatment with ATR inhibitors or other DDR related inhibitors (except poly ADP ribose polymerase enzyme (PARP) inhibitors)
4. Subjects with a history of another primary malignancy other than:

   1. carcinomas in situ, (e.g., breast, cervix, and prostate)
   2. Locally excised non-melanoma skin cancer
   3. No evidence of disease from another primary cancer for two or more years and has not taken any anti-cancer treatment in two years. Exceptions are gonadotropin-releasing hormone (GnRH) therapy for prostate cancer and hormonal maintenance therapy for breast cancer.
5. Previously received treatment with strong CYP3A4, CYP2C8 and P-gp inhibitors or strong CYP3A4, CYP2C8 and P-gp inducers within 14 days prior to the first medication
6. Patients with AE due to previous anti-tumor treatment that has not recovered to ≤ CTCAE grade 1 (except for alopecia, pigmentation and lymphopenia)
7. Patients who are unable to swallow the tablets normally, or have abnormal gastrointestinal function that may affect the drug absorption, such as malabsorption syndrome or major resection of the stomach or bowels based on the judgment of the investigator
8. Subjects with any severe and/or uncontrolled disease, including:

   1. Poor blood pressure control (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg)
   2. Myocardial infarction, arrhythmia (CTCAE grade 2 and above, also including ≥ Class II congestive heart failure (CHF) (New York Heart Association (NYHA) classification) (refer to Appendix-A)
   3. Active infection or fever of unknown origin ≥ 38.5℃ within 7 days prior to the first medication
   4. Active viral hepatitis; positive hepatitis B surface antigen and/or hepatitis B core antibody and measured HBV DNA value ≥ 500 IU/ml; positive HCV antibody and measured HCV titer exceeding the upper limit of normal;
   5. Positive Treponema pallidum antibody;
   6. History of immunodeficiency, including positive HIV antibody or other acquired or congenital immunodeficiency diseases, or history of organ transplant;
   7. Poor control of diabetes (fasting blood glucose (FBG) > 10 mmol/L);
   8. Liver disease such as decompensated liver disease
9. Uncontrolled pleural effusion, pericardial effusion, or peritoneal effusion as per the investigator opinion
10. Patients with clinically significant hemorrhage symptoms or bleeding tendency within 3 months prior to the first study medication
11. Known hypersensitivity or contraindication to any drug or any of the components of investigational product
12. Any other clinically significant acute or chronic medical or psychiatric or any laboratory abnormality that may increase the risk associated with study drug administration or may interfere with the interpretation of study results

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Phase I: To determine dose-limiting toxicity (DLT) at each dose level and identify MTD and RP2D. | 21 days
  Phase I: Dose Escalation To observe the tolerability and safety of TCC1727 tablets and determine the maximum-tolerated dose (MTD) and the recommended phase II dose (RP2D) of TCC1727 tablets when administered orally once a day (QD) in 21-day cycle in patients with advanced solid tumors.
Phase II: To evaluate the preliminary efficacy of TCC1727 tablets as measured by ORR in patients with advanced solid tumors with DNA damage response (DDR) defects | 6 months
  Phase II: Cohort Expansion ORR according to Response Evaluation Criteria in Solid Tumors (RECIST) guidelines (version 1.1, 2009) for each tumor type. The overall response rate is defined as proportion of subjects who had the best overall response (BOR) of complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Phase I: Dose Escalation To observe the preliminary efficacy of TCC1727 tablets as measured by overall response rate (ORR) in patients with advanced solid tumors. | 6 months
  To evaluate the preliminary efficacy by objective response rate (ORR), disease control rate (DCR), duration of response (DOR), progression free survival (PFS) and overall survival (OS).
Phase I: To evaluate the pharmacokinetic (PK) of TCC1727 tablets in patients with advanced solid tumors | 21 days
  Phase I: Dose Escalation Pharmacokinetic parameters: Tmax
Phase I: | 21 days
  Phase I: Dose Escalation Pharmacokinetic parameters: Cmax
Phase I: | 21 days
  Phase I: Dose Escalation Pharmacokinetic parameters: t1/2
Phase I: | 21 days
  Phase I: Dose Escalation Pharmacokinetic parameters: AUC0-t,
Phase I: | 21 days
  Phase I: Dose Escalation Pharmacokinetic parameters: Cmax,ss
Phase I: | 21 days
  Phase I: Dose Escalation Pharmacokinetic parameters: AUCtau,ss,
Phase I: | 21 days
  Phase I: Dose Escalation Pharmacokinetic parameters: Cmin,ss
Phase II: To evaluate the safety and tolerability of TCC1727 tablets in patients with advanced solid tumors with DDR defects | 6 months
  Phase II: Cohort Expansion Assessment of all AEs, SAEs and TEAEs;

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No